CLINICAL TRIAL: NCT04969406
Title: A Prospective Trial Designed to Evaluate the Repeatability and Reproducibility of the Intelon BOSS(TM) System
Brief Title: A Prospective Trial of the Intelon BOSS(TM) System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment Difficulty
Sponsor: Intelon Optics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P21-02
Record Dates: First submitted 2021-07-07; First posted 2021-07-20 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-03

CONDITIONS: Cornea; Lens Diseases
MeSH Terms: conditions — Corneal Diseases; Lens Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging by BOSS System (Experimental): Imaging by the BOSS System
  Interventions: Other: Brillouin Spectroscopy via BOSS System

INTERVENTIONS:
Other: Brillouin Spectroscopy via BOSS System — Biomechanical Imaging of the Cornea and Lens

SUMMARY:
A prospective, open-label, single-site clinical trial designed to evaluate the repeatability and reproducibility of biomechanical imaging by the BOSS device. Subjects will undergo unilateral biomechanical mapping of the cornea and lens by three BOSS devices operated by three (3) different operators.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Availability, willingness and sufficient cognitive awareness to comply with the examination procedures and schedule
3. Signed Written Informed Consent

Exclusion Criteria:

1. No light perception or low vision rendering the subject unable to fixate to keep gaze still enough to acquire images
2. Presence of corneal opacity
3. Presence of cortical cataracts visible in an undilated pupil
4. Any systemic disease or disorder which would prohibit image acquisition (e.g., Parkinson's Disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-07-24 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Analysis of variance in corneal and lens measurements to determine repeatability and reproducibility | Evaluation Visit (within 30 days of the Screening Visit)
  A random effect model will be used to assess variation due to device/operator configuration

CONTACTS AND LOCATIONS:
Locations (1):
- Vold Vision plc, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No